CLINICAL TRIAL: NCT02128997
Title: Prophylactic Wound VACuum Therapy to Decrease Rates of Cesarean Section in the Obese Population
Acronym: PROVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 819579
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Wound Complication
Keywords: obesity, cesarean section, wound complication
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Incision Wound vacuum (Prevena) (Experimental): Closed incision wound vacuum (Prevena)
  Interventions: Device: Closed incision wound vacuum (Prevena)
- Routine Wound Care (No Intervention): This arm includes patients having a cesarean section with routine wound care

INTERVENTIONS:
Device: Closed incision wound vacuum (Prevena) — wound vacuum to be placed on a closed incision
  Arms: Closed Incision Wound vacuum (Prevena)

SUMMARY:
This study will assess whether a negative pressure wound vacuum therapy (NPWT) on closed incisions decreases the risk of wound complications among obese patients after cesarean section

All patients having a cesarean section in labor or presenting to the triage unit and requiring a cesarean section will be eligible

Main study intervention: this involves the use of a negative pressure wound vacuum therapy on a closed incision.

DETAILED DESCRIPTION:
Objectives To evaluate whether there is a decrease in wound complications among obese patients who are treated with closed incision NPWT versus standard post cesarean section wound care protocol.

Primary outcome variable(s) The primary outcome variable is wound complications defined as any readmission for a wound issue within four weeks of discharge, infection, or wound breakdown.

Secondary outcome will look at patient quality of life among those with NPWT versus usual care arm.

A survey addressing pain, breast feeding questions and ability to perform activity of daily living will be administered during the inpatient stay and at the postpartum visit.

Background Obesity, defined as a body mass index (BMI) 30kg/m2, continues to be a growing epidemic in the United States. According to National Center for Health Statistics Data1, almost one third of adults and 17% of youth were obese in 2009-2010. Furthermore, non-Hispanic Blacks have the age-adjusted rates of obesity (49.5%). In a study by Chu et al analyzing data from 26 states in the Pregnancy Risk Assessment Monitoring System (PRAMS) database, 20% of women who delivered were obese and in certain ethnic and insurance subgroups, the rates were as high as 33%. In 2008, according to reports by the Pennsylvania State statistics, the rates of obesity in the city of Philadelphia were as high as 64%. Multiple studies have demonstrated the increased risks for diabetes, hypertension and adverse pregnancy outcomes (APO) during pregnancy in the obese population. In addition, obesity is a well established independent risk factor for the development of a wound complication or infection after a cesarean delivery, with rates ranging from 10-15% . Certain measures such as antibiotic prophylaxis and closure of the subcutaneous space are techniques that have demonstrated a decreased incidence of wound disruption. Currently no randomized controlled trials have looked at the effects of surgical approach or choice of abdominal incision in the obese or extremely obese woman undergoing cesarean delivery. However, the few retrospective studies that have addressed this issue have demonstrated mixed results. Given the paucity of randomized controlled trials evaluating the prevention of wound complications in obese women undergoing cesarean delivery, a recent review by Tipton emphasized the necessity for such trials to evaluate methods with which to improve postoperative wound care and healing in this high risk cohort. In the past decade, negative pressure wound therapy (NPWT) has become accepted in the treatment of expediting healing of open wounds 15-18. NPWT is a method in which a vacuum device is placed on the wound in order to remove excess interstitial fluid, increase tissue vascularity, decrease bacterial colonization, and place mechanical stress on adjacent wound edges which aids in wound contractility and closure. Therefore, the positive effects of NPWT on open wounds have been well studied and established. Recent studies have been performed to assess a potential effect of NPWT on closed incisions non-obstetric fields. A recent study by Grauhan et al compared the effects of NPWT over closed sternotomy incisions in obese patients compared to conventional sterile wound dressing and noted a significant reduction in the rates of wound infection in those treated with NPWT.

Another study by Vargo assessed the effects of NPWT on closed incisions in patients undergoing abdominal therapy compared to a historical control also noted a decreased wound infection rate and no evidence of skin necrosis. In contrast, a recent study by Masden et al. looked at rates of infection and dehiscence in patients with multiple comorbidities status post predominantly lower extremity wounds and did not appreciate a difference between the NPWT group and dry dressing group24. Therefore, the need for further studies assessing the benefits of NPWT on various anatomical sites has been clearly established.

ELIGIBILITY:
Key inclusion criteria BMI greater than or equal to 30 kg/m2 at less than or equal to 22 weeks of gestation Subject is laboring Subject is having an unplanned cesarean section Subject will have Pfannenstiel Skin Incision Subject has the ability to take a picture and email it to a secure account Subject receives prenatal care in the University of Pennsylvania health system and plans to follow up postpartum in the system Subject is greater than or equal to 18 years of age

Key exclusion criteria Subject cannot read or speak English Subject is not 18 years of age Subject does not have ability to send a picture by email Subject has preexisting diabetes mellitus (Type 1 or Type 2) , is using chronic steroids or immune-suppressants, OR being actively treated for a malignancy Subject is undergoing a scheduled cesarean section Subject is allergic to silver

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Durnwald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ruhstaller K, Downes KL, Chandrasekaran S, Srinivas S, Durnwald C. Prophylactic Wound Vacuum Therapy after Cesarean Section to Prevent Wound Complications in the Obese Population: A Randomized Controlled Trial (the ProVac Study). Am J Perinatol. 2017 Sep;34(11):1125-1130. doi: 10.1055/s-0037-1604161. Epub 2017 Jul 13. PMID 28704847

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
Started | 67 | 69
Completed | 61 | 58
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Continuous [Median (Standard Deviation); unit: Years] — Population: This population only includes patients who were not lost to follow up.
  Years
    number analyzed (Participants) | 58 | 58 | 116
    (all) | 27 (5) | 29 (3) | 28 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This population only includes patients who were not lost to follow up.
  Participants
    number analyzed (Participants) | 61 | 58 | 119
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 46 | 45 | 91
    White | 14 | 12 | 26
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 67 | 69 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Complications
Description: The primary outcome variable was a composite of wound morbidity at 4 weeks postpartum including SSI and/or wound opening
Time Frame: Four weeks after cesarean section
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
Number analyzed (Participants) | 61 | 58
Participants | 3 | 4

2. Secondary Outcome: Pain Scores
Description: On postoperative day 2, all patients were administered a pain scale: Rank sharp pain (0-10), 10 being worst possible sharp pain.
Time Frame: Postpartum day 2
Measure: Median (Inter-Quartile Range); unit: Unit on a scale
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
Number analyzed (Participants) | 61 | 58
Unit on a scale | 6 [4 to 8] | 5.5 [3 to 8]

3. Secondary Outcome: Tingling Pain Scores
Description: On postoperative day 2, all patients were administered a pain scale: Rank tingling pain (0-10), 10 being worst possible tingling pain
Time Frame: Postpartum day 2
Measure: Median (Inter-Quartile Range); unit: Unit on a scale
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
Number analyzed (Participants) | 61 | 58
Unit on a scale | 2 [0 to 6] | 1.5 [0 to 6]

4. Secondary Outcome: Postpartum Length of Stay
Time Frame: Until hospital discharge and then for 4 weeks follow up
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
Number analyzed (Participants) | 61 | 58
days | 3 [3 to 4] | 3 [3 to 4]

ADVERSE EVENTS:
Time Frame: 4 week followup
Arm/Group | Closed Incision Wound Vacuum (Prevena) | Routine Wound Care
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No